CLINICAL TRIAL: NCT06519552
Title: A Clinical Study Evaluating the Safety, Tolerability, and Initial Efficacy of JWK008 Given by a Single Intravenous Infusion in Patients With Mucopolysaccharidosis Type I
Brief Title: A Clinical Study Evaluating the Safety, Tolerability, and Initial Efficacy of JWK008 in Patients With Mucopolysaccharidosis Type I
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1287
Record Dates: First submitted 2024-06-23; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Mucopolysaccharidosis Type I
Keywords: Mucopolysaccharidosis Type I; MPS I; Gene Therapy; AAV; Adeno-associated virus
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWK008 injection (Experimental): The participants will be given 5.0×10^12vg/kg or 2.0×10^13vg/kg body weight of JWK008
  Interventions: Genetic: JWK008 Single intravenous infusion administration

INTERVENTIONS:
Genetic: JWK008 Single intravenous infusion administration — Six participants with MPS I will be enrolled in the study. The participantss will be divided into two different dose groups, and a "3+3" dose escalation design is used. The low dose is 5.0×10^12vg/kg, and the high dose is 2.0×10^13vg/kg. Only one intravenous infusion of JWK008 will be administered to each participant.

SUMMARY:
This study is a single-center, single-arm, non-randomized, open-label, non controlled, dose-escalation, prospective clinical trial designed to assess the safety, tolerability, and preliminary efficacy of JWK008 injection in patients with MPS I.

DETAILED DESCRIPTION:
MPS I is a rare autosomal recessive disease caused by deﬁciency of the α-L-iduronidase (IDUA) gene, which encodes a lysosomal enzyme required for degradation of glycosaminoglycans (GAGs).While currently available therapies, enzyme replacement therapy (ERT) and hematopoietic stem cell transplantation (HSCT), provide clinical benefit over untreated disease progression,they still have significant limitations. ERT does not cross the blood-brain barrier and, therefore, does not treat the central nervous system (CNS) effects of the disease. And HSCT, although it can prevent cognitive decline in patients, has a high mortality rate and morbidity. The investigators have designed a novel IDUA fusion protein with the ability to cross the blood-brain barrier through the addition of the brain-targeting peptide Mtfp. On this basis, the investigators constructed an IDUA gene expression cassette for liver-targeted expression, and used a highly efficient liver-specific promoter to make the IDUA gene specifically and efficiently expressed in liver tissue, and the expressed protein can enter the central nervous system to exert therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old;
2. Diagnosis of MPS type I;
3. Be able to understand the purpose, content, and possible risks of this clinical study, voluntarily participate in and sign the informed consent form;
4. If the subject is female, her sexual partner must agree to use reliable contraception until 2 consecutive tests of vector sequence in the blood are negative; If the subject is male, the subject agrees to use reliable contraception until the semen sample is negative for 2 consecutive tests of the vector sequence.
5. Magnetic resonance imaging (MRI) of the liver mass read by the radiologist is negative.

Exclusion Criteria:

1. Known to be unresponsive to ERT; or those who have been treated with intrathecal or intravenous laronidase and have serious adverse reactions, such as significant infusion-related reactions (IARs) or anaphylactic shock.
2. Serum AAV5 neutralizing antibody titer is greater than 1:100.
3. Has contraindications for Corticosteroids.
4. Current treatment with systemic (intravenous or oral) immunomodulators or steroid use (topical treatments such as asthma or eczema are allowed).
5. Has contraindications for lumbar puncture.
6. When filtering, one of the following situations exists:

   1. Hepatitis B surface antigen (HBsAg) is positive, and the copy number of hepatitis B virus deoxyribonucleic acid (HBV-DNA) is>the upper limit of normal value (ULN);
   2. Hepatitis C virus antibody (HCV-Ab) is positive, and the copy number of hepatitis C virus ribonucleic acid (HCV-RNA) is>ULN;
   3. Receiving antiviral treatment for hepatitis B or C;
   4. The human immunodeficiency virus (HIV) test is positive and the CD4+T lymphocyte count is ≤ 200/mm3;
7. Abnormal laboratory values considered clinically significant (ALT and/or AST >3× upper limit of normal (ULN), total bilirubin > 1.5× ULN, serum creatinine > 1.5× ULN, etc.).
8. Have a history of chronic infections or other chronic diseases that researchers believe pose an unacceptable risk;
9. Active severe infection or any other significant accompanying, uncontrolled medical condition(except for those caused by MPS I), including but not limited to kidney, liver, blood, gastrointestinal, endocrine, lung, nervous system, brain or mental illness, alcoholism, drug dependence, or any psychological disorder assessed by the researcher that may interfere with adherence to experimental protocol procedures or tolerance to JWK008 injection;
10. History of active malignancy within the past 5 years (non-melanotic skin cancer or carcinoma in situ of the cervix is allowed).
11. Circulating alpha-fetoprotein (AFP) is elevated or abnormal.
12. Previously received gene therapy or participated in interventional clinical studies within the past 12 weeks;
13. Pregnant or lactating females.
14. The researcher believes that the subject is not suitable to participate in any concurrent clinically significant major diseases or other situations in the study;
15. Unable or unwilling to comply with the visit and study evaluation schedule described in the clinical protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2026-06-22 (Estimated); Study Completion 2029-06-22 (Estimated)

PRIMARY OUTCOMES:
adverse events | 5 years
  Adverse events defined as the number of participants with adverse events according CTCAE 5.0

SECONDARY OUTCOMES:
IDUA enzyme activity in blood and cerebrospinal fluid | 5 years
  Changes in IDUA activity in blood and cerebrospinal fluid before and after treatment are detected by laboratory testing.
GAG levels in blood, urine, and cerebrospinal fluid | 5 years
  Changes in GAG levels in blood, urine, and cerebrospinal fluid before and after treatment are detected by laboratory testing.
Six-Minute Walk Test | 5 years
  The distance that the patient could withstand the fastest walking distance on flat ground within 6 minutes before and after treatment was measured
Range of the joint motion(JROM) testing by measuring ruler | 5 years
  A measuring ruler was used to detect changes in the participant's range of the joint motion before and after treatment
Liver and spleen size were detected by CT | 5 years
  Changes in liver and spleen size were detected by CT
Vector shedding | 5 years
  As measured by vector concentration (quantitative polymerase chain reaction to JWK008 deoxyribonucleic acid ) in CSF, serum, and urine

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Ph.D, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan Universit, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No